CLINICAL TRIAL: NCT00085462
Title: Treatment of Patients With Metastatic Melanoma by Lymphodepleting Conditioning Followed by Infusion of TCR-Gene Engineered Lymphocytes and Subsequent Fowlpox gp100 Vaccination
Brief Title: Gene-Modified White Blood Cells Followed By Interleukin-2 and Vaccine Therapy in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 040181; 04-C-0181; NCI-6470; CDR0000370798; NCT00082264 (obsolete NCT alias)
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Melanoma (Skin)
Keywords: recurrent melanoma; stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — aldesleukin; Filgrastim; Cyclophosphamide; fludarabine phosphate

INTERVENTIONS:
Biological: aldesleukin
Biological: filgrastim
Biological: gp100-fowlpox vaccine
Biological: therapeutic autologous lymphocytes
Biological: therapeutic tumor infiltrating lymphocytes
Drug: cyclophosphamide
Drug: fludarabine phosphate

SUMMARY:
RATIONALE: Inserting a gene that has been created in the laboratory into a person's white blood cells may make the body build an immune response to kill tumor cells. Interleukin-2 may stimulate a person's white blood cells to kill tumor cells. Vaccines may make the body build an immune response to kill tumor cells. Combining gene-modified white blood cell infusions with interleukin-2 and vaccine therapy may kill more tumor cells.

PURPOSE: This phase I trial is studying how well giving gene-modified white blood cells when given together with interleukin-2 and vaccine therapy works in treating patients with metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine, preliminarily, any clinical tumor regression in lymphodepleted patients with metastatic melanoma treated with fowlpox gp100 antigen immunization and antitumor antigen T-cell receptor (TCR)-engineered tumor infiltrating lymphocytes or CD8+ autologous peripheral blood lymphocytes followed by interleukin-2.

Secondary

* Determine the in vivo survival of TCR gene-engineered cells in patients treated with this regimen.

OUTLINE: Patients are stratified according to their ability to produce tumor-infiltrating lymphocytes (TIL) (yes vs no).

Patients receive lymphodepleting chemotherapy comprising cyclophosphamide IV over 1 hour on days -7 and -6 and fludarabine IV over 30 minutes on days -5 to -1.

* Stratum 1 (TIL): Patients receive TIL retrovirally transduced with gp100 antigen TCR gene IV over 20-30 minutes on day 0*.
* Stratum 2 (CD8+peripheral blood lymphocytes [PBL]): Patients receive CD8+PBL retrovirally transduced with gp100 antigen TCR gene IV over 20-30 minutes on day 0*.

NOTE: *Day 0 is 1-4 days after the last dose of fludarabine.

Patients in both strata also receive fowlpox-gp100 vaccine (before TIL/PBL infusion) IV over 1-2 minutes on days 0 and 28 and high-dose interleukin-2 (IL-2) IV over 15 minutes every 8 hours on days 0-4 and days 28-32. Patients also receive G-CSF SC once daily beginning on day 0 and continuing until blood counts recover.

Treatment continues in the absence of disease progression or unacceptable toxicity. Beginning 6-8 weeks after the last dose of vaccine and high-dose IL-2, patients with stable or responding disease may receive 1 retreatment course.

Responding patients are followed at 1, 3, 6, and 12 months and then annually thereafter.

PROJECTED ACCRUAL: A total of 61 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of melanoma

  * Metastatic disease
* Measurable disease
* Refractory to standard therapy, including high-dose interleukin-2 therapy
* HLA-A*0201 positive
* Progressive disease during prior immunization to melanoma antigens OR prior treatment with anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody (MDX-010) cellular therapy with or without myeloablation allowed provided toxicity resolved to ≤ grade 2 (except vitiligo) AND patient does not require systemic steroids
* No brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* More than 3 months

Hematopoietic

* Absolute neutrophil count > 1,000/mm^3
* Platelet count > 100,000/mm^3
* Hemoglobin > 8.0 g/dL
* Lymphocyte count > 500/mm^3
* WBC > 3,000/mm^3
* No coagulation disorders

Hepatic

* AST and ALT < 3 times upper limit of normal (ULN)
* Bilirubin ≤ 2.0 mg/dL (3.0 mg/dL in patients with Gilbert's syndrome)
* Hepatitis B surface antigen negative
* Hepatitis C antibody negative (unless antigen negative)

Renal

* Creatinine ≤ 1.6 mg/dL

Cardiovascular

* LVEF ≥ 45% by cardiac stress test

  * No LVEF < 45% in patients ≥ 50 years of age
* No myocardial infarction
* No cardiac arrhythmias
* No symptomatic cardiac ischemia
* No prior EKG abnormalities
* No other major cardiovascular illness

Pulmonary

* FEV_1 ≥ 60% of predicted AND no obstructive or restrictive pulmonary disease
* No symptoms of respiratory dysfunction
* No other major respiratory illness

Immunologic

* HIV negative
* Epstein-Barr virus positive
* No active systemic infections (including opportunistic infections)
* No form of primary (e.g., autoimmune colitis or Crohn's disease) or secondary immunodeficiency (due to chemotherapy or radiotherapy)
* No prior severe immediate hypersensitivity reaction to any of the study agents including eggs
* No other major illness of the immune system

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 4 month after study participation
* Willing to complete a durable power of attorney (DPA)

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* More than 6 weeks since prior MDX-010

Chemotherapy

* Not specified

Endocrine therapy

* See Disease Characteristics
* No concurrent systemic steroid therapy

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* More than 4 weeks since other prior systemic therapy and recovered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2004-05; Primary Completion 2007-05 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Rosenberg, MD, PhD, Principal Investigator — NCI - Surgery Branch
Locations (2):
- United States (2):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland
  - NCI - Surgery Branch, Bethesda, Maryland